CLINICAL TRIAL: NCT01433003
Title: The Plasma Large-Volume Exchange Randomized Controlled Trial (PLEX-RCT)
Brief Title: The Plasma Large-Volume Exchange RCT
Acronym: PLEX-RCT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr William F Clark, Professor, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 259509
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Purpura, Thrombotic Thrombocytopenic; Hemolytic Uremic Syndrome
Keywords: Thrombotic thrombocytopenia purpura; hemolytic uremic syndrome; plasma exchange; Improve treatment response; TTP/HUS
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Hemolytic-Uremic Syndrome | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard-dose plasma exchange (Active Comparator): 50-75 ml/kg/day
  Interventions: Procedure: Plasma Exchange
- High-dose Plasma Exchange (Experimental): 125 ml/kg/day up to 10 L/day
  Interventions: Procedure: Plasma Exchange

INTERVENTIONS:
Procedure: Plasma Exchange — Plasma exchange is a blood purification technique that removes plasma from the blood and replaces it with donor plasma.

SUMMARY:
Thrombotic thrombocytopenia purpura / hemolytic uremic syndrome (TTP/HUS) is a rare, life-threatening disorder. TTP/HUS causes multiple blood clots to form, which prevents blood from reaching the brain and kidneys. TTP/HUS affects 3-5 people per million per year. Anyone can develop TTP/HUS, but it is most common among 30-40 year olds, and women are twice as likely as men to acquire the condition. TTP/HUS sometimes develops as a result of medication use, pregnancy or cancer; however, for the majority of patients (80%) the cause of TTP/HUS is unknown. In 1991, researchers discovered that plasma exchange was superior to plasma infusion in treating idiopathic TTP/HUS. During plasma exchange the patient's blood plasma is removed and replaced with healthy blood plasma. Without plasma exchange, the survival rate for TTP/HUS is extremely low, with fewer than 5% of patients surviving. Treating TTP/HUS with plasma exchange improved the survival rate to 80%. Although this represents a dramatic improvement, researchers are still searching for methods to improve survival. No major advances in treating TTP/HUS have occurred in the past 20 years. Recent research suggests that high-dose plasma exchange may improve the survival of TTP/HUS patients. The investigators will conduct a randomized controlled trial to test whether treating TTP/HUS patients with high-dose versus standard-dose plasma exchange improves the treatment response. The investigators will recruit 150 patients with TTP/HUS from 9 centres across Canada over three years. The investigators will evaluate whether high-dose plasma exchange improves the treatment response, survival, and whether it reduces the number and volume of plasma exchange procedures and duration of hospital stay.

DETAILED DESCRIPTION:
Background: Thrombotic thrombocytopenia purpura / haemolytic uremic syndrome (TTP/HUS) is a rare blood disorder with a high mortality rate of >95% when left untreated. In 1991, researchers discovered that treating TTP/HUS with plasma exchange vs. plasma infusion dramatically improved the survival rate, from 60% to 80%.The optimal plasma dose for treating TTP/HUS is unknown; however, recent research suggests that high-dose plasma exchange may improve survival in patients with TTP/HUS.

Hypothesis: Treatment of TTP/HUS with high-dose vs. standard-dose plasma exchange will significantly decrease the composite outcome of 1) treatment failure at day 5 and/or 2) non-response or death at 2 weeks.

Methods: The investigators will conduct a multi-centre, parallel group randomized controlled trial. The investigators anticipate recruiting 150 eligible patients with idiopathic TTP/HUS from 9 centres across Canada over 2.25 years. Patients will be randomized to receive high-dose plasma exchange (125 ml/kg/day up to 10 L/day plasma volume) or standard-dose plasma exchange (50-75 ml/kg/day; approximately 1-1.5 plasma volume). The primary composite outcome includes treatment failure at day 5 or non-response or death from any cause at 2 weeks. Secondary outcomes include the individual components of the primary outcome, non-response or death from any cause at month 1 and month 6, days to remission, duration of hospital stay, number and volume of plasma exchange treatments, and cost minimization.

Research Team: Our multi-centre team is part of the Canadian Apheresis Group, which was established in 1980 and currently operates in 30 centres across Canada. Collectively, the Canadian Apheresis Group treats 150 TTP/HUS patients each year. Our team includes experienced haematologists, nephrologists, epidemiologists and a biostatistician. The investigators have successfully collaborated on several projects and have an excellent publication record (>50 publications across more than 15 journals including the New England Journal of Medicine).

Timeline and Budget: Because TTP/HUS is a relatively rare disorder (an orphan disease), the investigators will recruit patients over 2.25 years from across Canada to achieve a sufficiently large sample size. A cost minimization study will be carried out in conjunction with the RCT to provide insight into potential costing.

Future Directions: If the investigators can demonstrate that high-dose plasma exchange significantly improves the primary outcome, the investigators will pursue a multi-national collaboration with American, Chinese and European Centres to investigate other important outcomes including optimal dosing, cost-effectiveness and survival.

Implications: This study has the potential to be the first major advancement in treating TTP/HUS in twenty years.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 year-old
2. First presentation of TTP/HUS
3. Meet all of the following diagnostic criteria:

   * Platelet count < 150 x 109 /L
   * Microangiopathic haemolytic anaemia (blood film with presence of red blood cell fragmentation)
   * LDH > 1.25 X the upper limits of normal
   * No alternative diagnosis

Exclusion Criteria:

1. Secondary TTP/HUS
2. Relapsing TTP/HUS
3. Hypersensitivity to blood product
4. Patient has received 2 or more plasma exchange treatment since symptom started over the last 1 week
5. Received medication, including cyclosporine, cyclophosphamide, rituximab for treatment of TTP/HUS
6. Other causes of thrombocytopenia than TTP/HUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
treatment failure at day 5 and/or 2) non-response or death at 2 weeks | baseline to two weeks
  LDH >1.25 x the upper limit of normal at Day 5 and <50% decrease from initial value, or Initial platelet count <50 x 109/L with <100% rise at Day 5, or Initial platelet count 50-99 x 109/L with <50% rise at Day 5, or Initial platelet count 100-150 x 109/L with Day 5 <150x 109/L, or LDH >1.25 x the upper limit of normal at 2 weeks, or Platelet count <150 x 109/L at 2 weeks, or Persistent or new neurological symptoms at 2 weeks

SECONDARY OUTCOMES:
All-cause mortality | 1 month; 6 months,
  all-cause mortality at 1-month and 6-months after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Central Facility, London, Ontario, Canada